CLINICAL TRIAL: NCT06354816
Title: VENLID: A Prospective, Randomized, Double-blind, Controlled Trial on the Application of a 10%-Lidocaine Spray Prior to the Insertion of a Peripheral Intra-venous Catheter in Female Adults
Brief Title: VENLID: The Application of a 10%-Lidocaine Spray Prior to the Insertion of a Peripheral Intra-venous Catheter in Female Adults
Acronym: VENLID
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: V 2.0, 07Feb2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: dominant/ Saline solution isotonic 0.9% NaCl - non-dominant/Xylocaine 10% pump spray (Experimental): Vessel at the dorsum manus: dominant/ placebo - non-dominant/ LA (Local anaesthesia)
  Forearm/cubita: dominant/ placebo - non dominant/ LA (Local anaesthesia)
  Interventions: Drug: Xylocaine 10% pump spray; Drug: Saline solution isotonic 0.9% NaCl
- B: non-dominant/ Saline solution isotonic 0.9% NaCl - dominant/ Xylocaine 10% pump spray (Experimental): Vessel at the dorsum manus: non-dominant/ placebo - dominant/ LA (Local anaesthesia)
  Forearm/cubita: non-dominant/ placebo - dominant/ LA (Local anaesthesia)
  Interventions: Drug: Xylocaine 10% pump spray; Drug: Saline solution isotonic 0.9% NaCl
- C: non-dominant/ Xylocaine 10% pump spray - dominant/ Saline solution isotonic 0.9% NaCl (Experimental): Vessel at the dorsum manus: non-dominant/ LA (Local anaesthesia)- dominant/ placebo
  Forearm/cubita: non-dominant/ LA (Local anaesthesia) - dominant/ placebo
  Interventions: Drug: Xylocaine 10% pump spray; Drug: Saline solution isotonic 0.9% NaCl
- D: dominant/ Xylocaine 10% pump spray - non-dominant/ Saline solution isotonic 0.9% NaCl (Experimental): Vessel at the dorsum manus: dominant/ LA (Local anaesthesia) - non-dominant/ placebo
  Forearm/cubita: dominant/ LA (Local anaesthesia) - non-dominant/ placebo
  Interventions: Drug: Xylocaine 10% pump spray; Drug: Saline solution isotonic 0.9% NaCl

INTERVENTIONS:
Drug: Xylocaine 10% pump spray — First volunteers will undergo insertion of PIVC into the vessel of dorsum manus; 2-10 hours later: All volunteers will undergo insertion of PIVC into the forearm/cubita. Lidocaine spray 10 % serves as a local anesthesia is applied with a dispenser dispensing 0.1ml per pulse on the area of the skin, where the insertion of the PIVC is planned.
  Exposure time is 2 min, timed with an hour glass; validated prior to the study by a stop watch. 0.5 ml (5 pulses) of 10% lidocaine spray (equals 50mg of lidocaine) are to be applied before insertion of a PIVC 18 Gauge.
  Other Names: Lidocaine 10% pump spray
Drug: Saline solution isotonic 0.9% NaCl — First volunteers will undergo insertion of PIVC into the vessel at dorsum manus; 2-10 hours later: All volunteers will undergo insertion of PIVC into the forearm/cubita. Physiological saline solution serves as a placebo and is applied with a dispenser dispensing 0.1ml per pulse on the area of the skin, where the insertion of the PIVC is planned.
  Exposure time is 2 min, timed with an hour glass; validated prior to the study by a stop watch. 0.5 ml (5 pulses) of 10% lidocaine spray (equals 50mg of lidocaine) are to be applied before insertion of a PIVC 18 Gauge.
  Other Names: physiological Saline solution 0.9% NaCl

SUMMARY:
Volunteers are invited to undergo 4 insertions of a peripheral intra-venous 18-gauge catheter (PIVC); 2 insertions at the the start of the study on the plantar side of the hand/vessel at the dorsum manus, 2 insertions after 2-10 hours into the forearm/cubita with and without application of a 10-% lidocaine spray (5 hubs of xylocaine 10%-pump spray; AstraZeneca BV, Zoetermeer, The Netherlands) prior to the insertion of the PIVC.

DETAILED DESCRIPTION:
Visit schedule:

Visit 1 Screening: Informed consent, Inclusion and exclusion criteria, Medical history, urine pregnancy test

Visit 2 Treatment Day1: PIVC vessel dorsum manus+ PIVC forearm/cubita

Treatment Day 1:

First, volunteers will undergo insertion of PIVC into the vessel at the dorsum manus; Volunteers are randomized in 4 groups, volunteers serve as there own controls

2-10 hours later: All volunteers will undergo insertion of PIVC into the forearm/cubita, volunteers serve as their own controls.

Clinical investigation procedures:

Lidocaine spray 10 % and the placebo, physiological saline solution, are filled in neutral brown glas bottles with a dispenser dispensing 0.1ml per pulse of the dispenser by the Pharmacy of the Konventhospital Bermherzige Brüder Linz, The operator and the volunteers are unaware which bottle contains the 10% lidocaine and which bottle the saline solution. 5 pulses of either lidocaine 10% or saline are applied to the site of the planned venipuncture (plantar side of the hand/vessel at the dorsum manus), an hourglass indicating the 2 min time is turned. The tourniquet is then loosened. After 2 minutes the tourniquet is tightened agained, desinfection is performed, another 30 sec is waited-timed by an hourglass-and the insertion of the PIVC is performed. The following PIVC will be used: BD Venflon Pro Safety, BD Vialon Material; 18G 1.3 x 32 mm; (Beckton Dickinson Therapy, Helsingborg, Sweden). To check for success of the insertion of the PIVC 5 ml of saline is injected; either way (success/failure) the PIVC is to be removed and the pain caused by PIVC rated by NRS is recorded. A pressure bandage will be applied and the volunteer is checked for well being and discharged at the principal investigator's discretion. Then the same procedure is repeated on the other extremity.

Description of Randomization:

4 randomization groups are defined per protocol. "Dominant" refers to the stronger hand/forearm.

* Group A: dominant/Placebo - non-dominant/LA
* Group B: non-dominant/Placebo - dominant/LA
* Group C: non-dominant/LA - dominant/Placebo
* Group D: dominant/LA - non-dominant/Placebo

On the treatment day the subinvestigator will obtain a card for each subject in which the treatment for each subject is specified. There are 40 cards and each card specifies the treatment protocol for a single subject. See attached document 2023-507859-29 Randimization cards.

Randomization is performed by a standard randomization program; groups are stratified by where (dominant vs. non-dominant extremity) the first PIVC will be inserted and whether LA or placebo is used at the first PIVC insertion resulting in 4 distinct groups.

No effect of order of dominant/non-dominant and placebo/LA is expected and thus in the main statistical analysis (see above) the randomization will not be taken into account. Nevertheless, an additional statistical analysis will be run as sensitivity analysis where the both randomization factors will be used as control variables in an ANOVA model.

Neither the subinvestigator nor the subjects will know what the content of the bottles are.

The plantar side of the hand and the forearm/cubita are randomized separately into the four groups A,B,C,D. Afterwards hand and arm are combined with each other.

Two separate block randomizations are forseen for the plantar side of the hand/vessel at the dorsum manus and for forearm/cubita via Software R version 4.2.2

Medication:

Lidocaine spray 10 % (Xylocaine 10% pump spray; AstraZeneca BV, Zoetermeer, The Netherlands) and the placebo, physiological saline solution (NaCl 0,9% 250ml Fresenius KABI), are filled in neutral brown glass bottles with a dispenser dispensing 0.1ml per pulse of the dispenser by the Pharmacy of the Konventhospital Barmherzige Brüder Linz on the basis of AMG.

Lidocaine spray 10 % (Xylocaine 10% pump spray) and the placebo (physiological saline solution NaCl 0,9%), are filled in neutral brown glass bottles. Four bottles (a,b,c,d) are prepared by the pharmacy. 2 bottles each are available. 2 bottles with label "a" and "b" for plantar side of hand/vessel at the dorsum manus and 2 bottles with label "c" and "d" for forearm/cubita. One of the bottles "a" and "b" is a placebo and the other one the local anaesthetic. One of the bottles "c" and "d" is a placebo and the other one the local anaesthetic.

The content of these bottles are only known by the Sponsor and the pharmacy.

The person responsible for PIVC insertion and the volunteers are unaware which bottle contains the 10% lidocaine and which bottle the saline solution. Due to the banana like smell of lidocaine the person responsible for PIVC insertion and the volunteer will wear nose clips during the procedure.

Null hypothesis:

There is no difference in pain with and without application of LA for the plantar side of the hand/vessel at the dorsum manus, and the forearm/cubita.

Alternative hypothesis:

There is a difference in pain with and without application of LA for the plantar side of the hand/vessel at the dorsum manus, and the forearm/cubita.

Primary objective:

• To demonstrate a reduction of pain caused by PIVC rated by Numerical Rating Scale (NRS), after application of a 10% lidocaine spray- Separately measured for the plantar side of the hand/vessel at the dorsum manus, and for the forearm/cubita.

Secondary objectives:

* To measure pain caused by PIVC rated by NRS in the dominant vs. non-dominant arm
* To measure pain caused by PIVC rated by NRS at the plantar side of the hand/vessel at the dorsum manus, vs. at the forearm/cubita
* To measure the correlation between pain caused by PIVC rated by NRS and the anticipated pain rated by NRS
* To measure the correlation between pain caused by PIVC rated by NRS and the anticipated difficulty by the operator to insert the PIVC
* To measure pain rated by NRS depending on success
* To describe success rates and compare it
* To measure the correlation between PCS and pain caused by PIVC rated by NRS

Statistics Pain caused by PIVC rated by NRS with/without application of local anesthesia will be analyzed by a paired- t-test. NRS is used as a continuous measure and we expect the values to be approximately normally distributed and therefore plan a parametric test. Normal distribution will be investigated via Q-Q-plots. If there is no normal distribution, the non-parametric Wilcoxon test for paired samples will be used instead of the paired t-test. For descriptive analyses, mean values and standard deviations will be reported. For each primary outcome (plantar side of the hand/vessel at the dorsum manus and the forearm) separate significance tests for separate null hypotheses will be calculated and no adaption of the error due to multiple testing is needed. The analysis will be performed with the SPSS software (SPSS 32.0, SPSS Inc., Chicago, IL).

For the analysis of the secondary endpoints paired t-test, independent t-tests and pearson correlation will be used. If the data is not normal distributed, wilcoxon test for paired samples, Mann-Whitney-U test for independent samples and spearman correlation will be employed instead. For analyzing the success rate a chi-squared test will be calculated for comparison of groups.

ELIGIBILITY:
Inclusion Criteria

* Female probands 18-45 years
* Personal history of ever having a venipuncture or insertion of PIVC

Exclusion Criteria

* Fractures on the upper extremity resulting in permanent movement restriction
* Significant burns on the upper extremity-at the discretion of the principal investgator
* Personal history of any thrombosis
* Personal history of chemotherapy
* Potential allergy to a PIVC
* Personal history of surgery in the axilla
* Personal history of any pathologies in the blood coagulation pathway
* Personal history of difficult peripheral venous access
* Personal history of complications with a PIVC
* Any concomitant use of an analgesic within the previous 24 h
* Any concomitant use of anticoagulation
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female volunteers
Enrollment: 40 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To demonstrate a reduction of pain caused by PIVC rated by Numerical Rating Scale (NRS), after application of a 10% lidocaine spray- Separately measured for the plantar side of the hand/vessel at the dorsum manus, and for the forearm/cubita | 2 minutes
  rated by a Numerical Rating Scale (NRS) from minimum 0 to maximum 10. Higher score means worse outcome

SECONDARY OUTCOMES:
To measure pain caused by PIVC rated by NRS in the dominant vs. non-dominant arm | 2 minutes
  rated by a Numerical Rating Scale (NRS) from minimum 0 to maximum 10. Higher score means worse outcome
To measure pain caused by PIVC rated by NRS at the plantar side of the hand/vessel at the dorsum manus vs. at the forearm/cubita | 2 minutes
  rated by a Numerical Rating Scale (NRS) from minimum 0 to maximum 10. Higher score means worse outcome
To measure the correlation between pain caused by PIVC rated by NRS and the anticipated pain rated by NRS | 2 minutes
  rated by a Numerical Rating Scale (NRS) from minimum 0 to maximum 10. Higher score means worse outcome
To measure the correlation between pain caused by PIVC rated by NRS and the anticipated difficulty by the operator to insert the PIVC | 2 minutes
  Injection of 5 ml physiological saline solution; 5. Success rate of the venipuncture by descriptive analysis and chi-square test for comparing success rate between hand and forearm.
To measure pain rated by NRS depending on success | 2 minutes
  rated by a Numerical Rating Scale (NRS) from minimum 0 to maximum 10. Higher score means worse outcome
To describe success rates and compare it | 2 minutes
  Injection of 5 ml physiological saline solution. Success rate of the venipuncture by descriptive analysis and chi-square test for comparing success rate between hand and forearm.
To measure the correlation between PCS and pain caused by PIVC rated by NRS | 2 minutes
  rated by a Numerical Rating Scale (NRS) from minimum 0 to maximum 10. Higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Hefler, MD, Principal Investigator — Depatment of Gynekology, Ordensklinikum Linz GmbH, Barmherzige Schwestern

IPD SHARING:
Plan to Share IPD: No